CLINICAL TRIAL: NCT02062294
Title: Retrospective Review of Valganciclovir Efficacy in Preventing CMV Disease in D+/R- Liver Transplant Recipients - A Non-Interventional Program
Brief Title: An Observational Study of Valcyte (Valganciclovir) in D+/R- Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25224
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective review will evaluate the efficacy of Valcyte (valganciclovir) in preventing Cytomegalovirus (CMV) disease in D+/R- liver transplant recipients. Data from eligible patients will be collected for the 6 months following transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients, >/= 16 years of age
* Transplantation between January 2004 and June 2009
* CMV seronegative recipient (R-) who received a liver transplant from a seropositive donor (D+)
* Valganciclovir therapy for at least 70 days beginning within 10 days post transplantation
* Assessment of CMV disease status within the first 6 months post transplantation

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplant recipients at high risk of developing Cytomegalovirus disease
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-07-31 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Switzerland (3):
  - Inselspital Bern; Viszerale Chirurgie und Medizin, Bern
  - HUG; Transplantation, Geneva
  - Universitätsspital Zürich; Klinik für Gastroenterologie und Hepatologie, Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 09 July 2010 and 22 September 2011 and recruited participants from 3 sites in Switzerland.
Pre-assignment Details: A total of 14 participants who were CMV seronegative and had received a liver transplant from a CMV seropositive donor, received 900 mg Valganciclovir in this study.
Groups:
- Valganciclovir: Each participant who received 900 mg Valganciclovir for at least 70 days beginning within 10 days post transplantation was observed.
Period: Overall Study
Arm/Group | Valganciclovir
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Valganciclovir
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 48 [17 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Developing Cytomegalovirus (CMV) Disease Within 6 Months of Liver Transplantation Under Valcyte Prophylaxis
Description: Participants with clinical manifestation of CMV disease within 6 months after liver transplantation under Valcyte prophylaxis were evaluated.
Time Frame: 6 months
Population: Per Protocol (PP) population comprised all 14 participants receiving Valganciclovir within 10 days post-transplantation for at least 70 days and for whom source data from the time period between liver transplantation until 6 months post-transplantation was available.
Measure: Number; unit: participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 14
participants | 3

2. Secondary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) or Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: 6 months
Population: Safety Analysis population (SAP) comprised all 14 participants which entered study.
Measure: Number; unit: participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 14
participants
  SAEs | 6
  AEs | 10

ADVERSE EVENTS:
Time Frame: 6 months
Description: Safety Analysis population (SAP) comprised all 14 participants which entered study.
Arm/Group | Valganciclovir
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir (N=14)
Incisional Hernia (Injury, poisoning and procedural complications) | 1
Transplant Rejection (Immune system disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cytomegalovirus Syndrome (Infections and infestations) | 2
Hepatitis C (Infections and infestations) | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir (N=14)
Abdominal pain (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Influenza like illness (General disorders) | 2
Oedema (General disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Cytomegalovirus syndrome (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Eye oedema (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.